CLINICAL TRIAL: NCT00408382
Title: Lipitor Phase 4 Clinical Trial in Hypercholesteremia Patients With Yellow Coronary Plaque
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5481/HOP1
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2006-12

CONDITIONS: Hypercholesteremia; Coronary Artery Disease
Keywords: Lipitor; atorvastatin; Hypercholesteremia; yellow coronary plaque
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin, Lipitor

SUMMARY:
To evaluate the efficacy of intensive lipid-lowering therapy with Lipitor on the changes of characteristics of yellow coronary plaque in subjects with hypercholesteremia accompanying coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypercholesteremia
* The indication of coronary angiography, coronary angioscopy and intravascular ultrasound are expected

Exclusion Criteria:

* Patients who has current administration of Lipitor or history of discontinued administration of Lipitor
* Acute cardiac infarction

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50

PRIMARY OUTCOMES:
Changes in plaque characteristics as observed by coronary angioscopy
(the amount of yellow plaque and grade shall be determined by the coronary angioscopic findings evaluation committee)
Changes in the volume and the echogenicity as observed by intravascular ultrasound

SECONDARY OUTCOMES:
Rate of change in serum lipid level
Changes in the surface character and size of plaque as observed by coronary angioscopy (determined by the angioscopic findings evaluation committee)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

REFERENCES:
- [Background] Hirayama A, Saito S, Ueda Y, Takayama T, Honye J, Komatsu S, Yamaguchi O, Li Y, Yajima J, Nanto S, Takazawa K, Kodama K. Qualitative and quantitative changes in coronary plaque associated with atorvastatin therapy. Circ J. 2009 Apr;73(4):718-25. doi: 10.1253/circj.cj-08-0755. Epub 2009 Feb 18. PMID 19225206